CLINICAL TRIAL: NCT01603355
Title: An Open-label Trial to Assess the Efficacy and Safety of Tocilizumab in the Management of Juvenile Idiopathic Arthritis Associated Vision-threatening Uveitis That is Refractory to Other Modes of Systemic Immunosuppression
Brief Title: Tocilizumab in the Management of Juvenile Idiopathic Arthritis Associated Uveitis
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: insufficient enrollment
Sponsor: Eric B. Suhler (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Eric B. Suhler, Principal Investigator, Oregon Health and Science University
Organization: Oregon Health and Science University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: e8343
Record Dates: First submitted 2012-05-18; First posted 2012-05-22 (Estimated); Results first posted 2018-11-27 (Actual); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Juvenile Idiopathic Arthritis Associated Uveitis
Keywords: JIA
MeSH Terms: interventions — tocilizumab

ARMS (1):
- Tocilizumab (Experimental)
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — Intravenous tocilizumab:
  Patients less than 30 kg weight:10 mg per kg every 4 weeks Patients at or above 30 kg weight: 8 mg per kg every 4 weeks
  Other Names: Actemra

SUMMARY:
The investigators are doing this research study to see if tocilizumab (Actemra) is safe and effective when used for severe or refractory non-infectious uveitis. Uveitis is an inflammation of the eye that is caused by the body's immune system reacting against the eye tissues.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with Juvenile Idiopathic Arthritis
* Subjects with vision-threatening autoimmune uveitis.
* Failure to respond to methotrexate or at least one other systemic immunosuppressive or intolerance to such medications due to side effects. Failure to respond includes presence of one plus or greater anterior chamber cell in both eyes; need for topical corticosteroid four times or more in either eye; ocular hypertension or glaucoma attributable to the topical corticosteroid.
* Subjects with bilateral disease.
* If subjects are on oral corticosteroids, the dosage must be stable for 2 weeks prior to baseline and not exceed 10 mg per day or 2mg/kg/day (whichever is less) of prednisone or its equivalent. Subjects must be willing to agree to not alter the dosage of oral steroids during the first 16 weeks of the trial.
* Must have a chest radiograph within 3 months prior to enrollment with no evidence of malignancy, infection or fibrosis.
* Parent or guardian must understand and voluntarily sign an informed consent form.
* Pediatric subjects of either gender 2-17 years at time of consent.

Exclusion Criteria:

* Inability of parent or guardian to provide voluntary consent
* Major surgery (including joint surgery) within 8 weeks prior to screening or planned surgery within 12 months following randomization.
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study
* Pregnant or breastfeeding
* Current liver disease, as determined by the Principal Investigator on the basis of history or serum studies
* History of severe allergic or anaphylactic reactions to human, humanized or murine monoclonal antibodies including tocilizumab.
* Evidence of significant uncontrolled concomitant diseases such as nervous system, renal, hepatic (patients with prior history of ALT elevation will not be excluded), endocrine, or gastrointestinal (GI) disorders, which in the Investigator's opinion, would preclude patient participation.
* Uncontrolled disease states, such as asthma, psoriasis or inflammatory bowel disease where flares are commonly treated with oral or parenteral corticosteroids.
* Any major episode of infection requiring hospitalization or treatment with IV antibiotics within 4 weeks of screening or oral antibiotics within 2 weeks prior to screening
* History of active mycobacterial infection with any species (including Mycobacterium tuberculosis) within 2 years prior to screening visit. Subjects with Mycobacterium tuberculosis infection more than 2 years prior to screening visit are allowed if successful treatment was completed at least 2 years prior to randomization and is documented and available for verification.
* Immunization with a live/attenuated vaccine within 4 weeks prior to baseline
* Latent Mycobacterium tuberculosis infection as indicated by a positive Purified Protein Derivative [PPD] skin test. Subjects with a positive PPD skin test and documented completion of treatment for latent TB are eligible. Subjects with a positive PPD skin test and not treated or no documentation of completion of treatment are ineligible.
* If QuantiFERON® test is performed instead of the PPD test, only those with a negative QuantiFERON® test are allowed in the study.
* History of incompletely treated Mycobacterium tuberculosis infection as indicated by

  * Subject's medical records documenting incomplete treatment for Mycobacterium tuberculosis
  * Subject's self-reported history of incomplete treatment for Mycobacterium tuberculosis
* History of recurrent bacterial infection (at least 3 major infections resulting in hospitalization and/or requiring intravenous antibiotic treatment within the past 2 years) or recurrent viral, fungal, mycobacterial, or other infections (including but not limited to atypical mycobacterial disease, hepatitis B and C, and herpes zoster, but excluding fungal infections of the nail beds)
* Clinically significant abnormality on the chest x-ray (CXR) at screening. Chest x-rays performed within 3 months prior to start of study drug are acceptable.
* Use of any investigational medication within 4 weeks prior to start of study drug or 5 pharmacokinetic/pharmacodynamic half-lives (whichever is longer)
* History of congenital or acquired immunodeficiency (eg, Common Variable Immunodeficiency [CVID])
* Hepatitis B surface antigen positive or Hepatitis B core antibody positive at screening
* History of Human Immunodeficiency Virus (HIV) infection
* Antibodies to Hepatitis C at screening
* Malignancy or history of malignancy (except for treated [ie, cured] basal-cell skin carcinomas > 3 years prior to screening)
* Have multiple sclerosis or other central demyelinating disorder.
* Presence of a transplanted organ (with the exception of a corneal transplant performed > 3 months prior to enrollment).
* History of substance abuse (drug or alcohol) within the previous 3 years, history of noncompliance to medical regimens, or other condition/circumstance that could interfere with the subject's adherence to protocol requirements.
* Previous or current use of an alkylating agent (e.g. chlorambucil or cyclophosphamide).
* Treatment with etoposide (VP16) within 3 months prior to the baseline visit.
* Administration of intravenous immunoglobulin for the treatment of active polyarticular disease within 4 weeks prior to the baseline visit.
* Previous treatment with any cell depleting therapies, including investigational agents (e.g. anti-CD19 and anti-CD20).
* Prior stem cell transplant at any time.
* TNF -blocker use within the 8-weeks prior to enrollment (Infliximab use within 10 weeks prior to enrollment).
* Laboratory Exclusion criteria (at screening):

  * Serum creatinine >1.5 ULN (upper limit of normal for age and sex);
  * AST or ALT > 1.5 ULN (upper limit of normal for age and sex);
  * Total bilirubin > 1.3 mg/dL (> 23 umol/L);
  * Platelet count < 150 x 103/μL (< 150,000/mm3);
  * Hemoglobin < 9.0 g/dL (< 3.7 mmol/L);
  * WBC count < 5,000/mm3 (< 5.0 x 109/L);
  * Neutrophil count < 2,500/ mm3 (< 2.5 x 109/L)

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2013-11; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric B Suhler, MD,MPH, Principal Investigator — Oregon Health and Science University; James T Rosenbaum, MD, Study Director — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tocilizumab
Started | 3
Completed | 1
Not Completed | 2
Not completed — Lack of Efficacy | 2

BASELINE CHARACTERISTICS:
Arm/Group | Tocilizumab
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 3
Participants with control of ocular inflammation at trace or less [Count of Participants; unit: Participants] | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Control of Ocular Inflammation
Description: control of anterior chamber cell in both eyes at week 16 to a level of trace or less (SUN criteria) without an increase in any immunosuppressive treatment and while using prednisolone acetate topically no more than 2 times per day
Time Frame: 16 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 3
Participants | 1

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Tocilizumab
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes